CLINICAL TRIAL: NCT05790135
Title: Evaluation of the Role of Multiparametric Ultrasound Study in Discriminating Among Intestinal Complications After Hematopoietic Stem Cell Transplantation. A Pilot Study.
Brief Title: Multiparametric Ultrasound Study in Diagnosing GvHD
Acronym: ECO-STEM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to enroll
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4926
Record Dates: First submitted 2023-03-07; First posted 2023-03-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Intestinal GVHD
Keywords: SCT; GvHD; gastrointestinal; CEUS; SWE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multiparametric ultrasound evaluation (Experimental): Multiparametric ultrasound evaluation will be applied to all patients who will develop diarrhea above 500 ml per day.
  Interventions: Device: shear wave elastography

INTERVENTIONS:
Device: shear wave elastography — Shear wave elastography and CEUS will be used to evaluate the reliability in diagnosing graft versus host disease of the gut after hematopoietic stem cell transplantation
  Other Names: contrast enhanced ultrasould (CEUS)

SUMMARY:
The study evaluate the role of the use of bed-side multiparametric ultrasound study in the diagnosis of gastrointestinal acute graft-versus host disease (aGvHD) in patients underwent allogenic stem cell transplantation

DETAILED DESCRIPTION:
The literature reports various experiences on the use of shear wave elastography (SWE) in the study of the intestine, especially in patients with chronic inflammatory bowel diseases. But few data are reported on the use of the method in patients with graft versus host disease. Considering the simplicity of the method, we think it can be applied to an ultrasound study of the intestine to try to understand the potential of SWE to further define the characteristics of the intestinal segments involved.

Study population will include all patients submitted to allogenic stem cell transplantation (SCT) who developed diarrhea > 500 ml per day suggestive for aGvHD until 100 days from transplant date. Patients submitted to autologous stem cell transplant who developed diarrhea between transplant date and engraftment achievement will constitute control population as for other infectious complications assessment. Within 24-48 hours from symptoms, onset full panel of stool cultures will be performed together with Clostridium toxin assessment. Multiparametric ultrasound study will be performed at the onset of the symptoms and then weekly to monitoring intestinal changes accordingly to symptoms evolution during treatment. In the case with high suspicion for aGvHD (stool culture negative, persistent or progressive diarrhea, ultrasound imaging closely suggestive for aGvHD), as per common clinical practice, colonoscopy will be required to evaluate internal macroscopy features of the bowel and to obtain histological samples for conclusive diagnosis. In the meantime steroid therapy will be started, as per common clinical practice. The only modification of this protocol to common clinical practice is represented by the addition of a non-invasive bed-side method of evaluation of the patients with diarrhea. None of the routinely performed diagnostic and therapeutic process will be modified. All patients submitted to autologous stem cell transplant who developed diarrhea between transplant date and engraftment achievement will constitute control population. Also in this case full panel of stool culture and clostridium toxin assessment will be performed at the onset of the symptoms. Multiparametric ultrasound study will be made al symptoms onset and then weekly until symptom resolution. Multiparametric ultrasound study will be performed by expert qualified staff as following:The examinations will be performed at patient's bed, in supine position, with a MyLab™9 Platform (by Esaote corporate, Italy) system. Fasting is required.

US for bowel requires both low-frequency convex probes (3.3-5 MHz) and high-frequency (5-17 MHz) linear assay probes to increase the spatial resolution of the intestinal wall and to assess the wall diameter and wall layer.

Primary endpoint of the study is to evaluate the accuracy of bed-side multiparametric ultrasound study in the diagnosis of gastrointestinal aGvHD in patients underwent to allogenic transplant in terms of sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV). Secondary endpoints To assess potential associations between bed-side multiparametric ultrasound measurements weekly performed and aGvHD diagnosis in patients underwent to allogenic transplant. To assess whether bed-side multiparametric ultrasound measurements at baseline differ in distinguishing complications different from aGvHD (i.e., infectious, drug-related o neutropenic colitis) in patients underwent allogenic transplant as compared to auto-transplant

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Submitted to first allogeneic stem cell transplant during the 12 months period of enrollment of the study;
* Diarrhea onset between day 0 and day +100 from transplant;
* Signed informed consent.

Exclusion Criteria:

* Previous allogeneic stem cell transplantation;
* Patients refusing to sign informed consent for the study;
* Patients affected by severe cardiomyopathy and respiratory distress/insufficiency;
* Patients unable to fully understand and accept study protocol for various problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of bed-side multiparametric ultrasound study in gut-GvHD diagnosis will be measured and reported | Onset of gastrointestinal symptoms within 100 days from transplant
  Primary endpoint of the study is to evaluate the sensitivity of bed-side multiparametric ultrasound study in the diagnosis of gastrointestinal aGvHD in patients underwent to allogenic transplant
Specificity of bed-side multiparametric ultrasound study in gut-GvHD diagnosis will be measured and reported | Onset of gastrointestinal symptoms within 100 days from transplant
  Primary endpoint of the study is to evaluate the specificity of bed-side multiparametric ultrasound study in the diagnosis of gastrointestinal aGvHD in patients underwent to allogenic transplant

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Metafuni, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT05790135/Prot_SAP_000.pdf